CLINICAL TRIAL: NCT06751823
Title: "Serum Zinc Levels and Intake in Type 2 Diabetes: Impact on Pathogenesis and Glycemic Control"
Brief Title: Evaluation of Zinc in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Heliopolis University (Other)
Responsible Party: Principal Investigator, Sara mostafa ElAdawy, lecturer, Heliopolis University
Other Study IDs: MD-81-2024
Record Dates: First submitted 2024-12-17; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
Keywords: type 2 DM,; zinc
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: haelthy volunteers
- Type 2 DM patients: patients of Type 2 DM with no known complications

SUMMARY:
investigation of the impact of zinc level on the development of DM and to elaborate on whether daily consumption of zinc affects the disease's evolution.

DETAILED DESCRIPTION:
The relationship between the pathophysiology of diabetes mellitus and trace element dysregulation emphasizes how crucial it is to maintain appropriate micronutrient status in order to manage this chronic metabolic disease. One promising strategy for enhancing glycemic control and lowering the risk of diabetic complications may be to address these underlying dietary imbalances.

Accordingly, the aim is to investigate the impact of zinc level on the development of DM and to elaborate on whether daily consumption of zinc affects the disease's evolution.

ELIGIBILITY:
Inclusion Criteria:

* confirmed Type 2 DM with no known complication
* more than or equal 40 years old

Exclusion Criteria:

pregnancy and lactation type 1DM known DM complication other endocrinological disorders malignancy

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: type 2 DM patients with no complication in comparison with health volunteers
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
zinc serum level in the participnats | "through study completion, an average of 1 year"
  investigate the impact of zinc serum level on the development of DM
Dietary micronutrient assessment using food questionnaire | "through study completion, an average of 1 year"
  Dietary micronutrient assessment using food questionnaire adopted from a questionnaire for screening the micronutrient intake of economically active South African adults
Trace elements daily intake calculation | "through study completion, an average of 1 year"
  It will be calculated by multiplying the element contents measured in food (μg/kg) with the intake as estimated by the food micronutrient questionnaire (g/day).
the dietary intake by kilogram (kg) of body weight (bw) | "through study completion, an average of 1 year"
  the dietary intake by kilograms (kg) of body weight (bw) by dividing by the weight of participants.

SECONDARY OUTCOMES:
HbA1C mesurements | "through study completion, an average of 1 year"
  investigate the impact of serum zinc level on the glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: sara eladwy, lecturer, Principal Investigator — Helioplis university
Locations (1):
- Cairo University Hospitsl, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be assigned codes with no needs to share IPD